CLINICAL TRIAL: NCT00315627
Title: Steroid-free and Long-term Calcineurin-free Trial in Islet Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rodolfo Alejandro (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0205
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Islet Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- islet transplantation (Experimental): Islet Alone Transplantation under Alentuzumab (Campath1H) induction.
  Interventions: Drug: Islet transplantation

INTERVENTIONS:
Drug: Islet transplantation — Islet transplantation
  Other Names: islet

SUMMARY:
The purposes of this study are:

1. To reverse hyperglycemia and insulin dependency in patients with type 1 diabetes mellitus through islet transplantation utilizing steroid free, calcineurin-inhibitor free immunosuppression.
2. To assess the long-term function of successful islet transplants in patients with type 1 diabetes mellitus utilizing islets that have undergone a period of culture.
3. To determine whether the natural history of the microvascular, macrovascular, and neuropathic complications are altered following the successful transplantation of islets.

DETAILED DESCRIPTION:
STUDY DESIGN:

The initial proposal submitted to the JDRFI was to compare 3 different groups of patients receiving islet cell transplants utilizing steroid-free, calcineurin-free protocols. The 3 groups were as follows:

1. Zenapax, Rapamycin & MMF
2. Campath, Rapamycin & MMF, and
3. Thymoglobulin, Rapamycin & MMF.

The grant was awarded in December 2003, however the recommendations were to focus on a single group (group 3 or 4) in order to determine the relative efficacy and toxicity of a new immunosuppressive drug combination. We elected to perform the group utilizing Campath, since we have a similar protocol utilizing the same immunosuppressive regimen with the addition of CD34+ enriched donor bone marrow cells (2000/0024). The results of this trial utilizing a steroid-free/calcineurin-free protocol will be compared with the standard "Edmonton Protocol" (2000/0196), which we are currently conducting (14 patients have been transplanted). In addition, the results will be compared with those in 2000/0024.

Protocol 2000/0024 (utilizing the same immunosuppressive regimen; Campath, Rapamycin, Tacrolimus-switched to MMF at 3 months) is being followed by a DSMB established at the NIH.

We propose to evaluate 12 patients with steroid free, long term calcineurin inhibitor free immunosuppression regimens which can be directly compared to our historical group of patients who underwent the Miami version of the Edmonton protocol (Islet Cell Transplantation Alone in Patients with Type 1 Diabetes Mellitus: Steroid-Free Immunosuppression - Protocol # 2000/196) and with the concurrent tolerogenic protocol (Islet Cell Transplantation Alone and CD34+ Enriched Donor Bone Marrow Cell Infusion in Patients with Type 1 Diabetes Mellitus; Steroid Free Regimen - Protocol # 2000/0024) which uses the same immunosuppressive regimen combined with CD34+ stem cell enriched donor bone marrow infusions.

The regimen will consist of Campath 1-H induction, maintenance immunosuppression with sirolimus and tacrolimus for 3 months with subsequent introduction of mycophenolate mofetil (MMF) and removal of tacrolimus completely and TNF-alpha inhibition (etanercept) in the peri-transplant period.

ELIGIBILITY:
Inclusion Criteria:

Potential candidates must have type 1 diabetes mellitus and fulfill one or more of the following:

1. Manifest signs and symptoms that are severe enough to be incapacitating. Incapacitating signs and symptoms include hypoglycemic episodes requiring assistance by others and hypoglycemia unawareness (the inability to recognize low blood glucoses; glucoses < 54 mg/dl). These patients are at high risk for involvement in accidents (they can lose consciousness or act irrationally), thus causing harm to themselves and/or others.
2. Patients with poor diabetes control (HbA1c > 8.0% but < 12%), despite intensive insulin therapy, as defined by: self monitoring of blood glucose ≥ 4 times/day, multiple insulin injections (≥ 3/day) or insulin pump, and close monitoring of blood glucose control by an endocrinologist. These patients can experience acute, rapid hyperglycemia secondary to several stress factors, that can lead to dehydration, disorientation, and in some instances, ketoacidosis.
3. Progressive diabetic complications. These patients with chronically poor glycemic control are at higher risk for the development of a wide variety of complications (retinopathy, neuropathy, nephropathy, and cardiovascular disease) associated with diabetes.

Exclusion Criteria:

Potential candidates will be excluded as per the following criteria:

1. Age < 18 or > 65 years
2. Duration of diabetes < 5 years
3. Do not have a physician that is monitoring diabetes for > 6 months
4. Body mass index > 26
5. Weight > 80 kg
6. Insulin requirement > 1.0 u/kg/d
7. HbA1c > 12%
8. Stimulated or basal C-peptide > 0.3 ng/ml
9. Corrected creatinine clearance < 60 ml/min
10. Serum creatinine consistently above 1.6 mg/dl
11. Macroalbuminuria (> 300 mg/24 hours)
12. Anemia (hemoglobin < 12.0 g/dl for males; < 11 g/dl for females)
13. Hyperlipidemia (fasting low-density lipoprotein [LDL] cholesterol > 130 mg/dl and/or fasting triglycerides > 200 mg/dl)
14. Abnormal liver function tests (consistently > 1.5 x normal range)
15. Serological evidence of HIV, HBsAg and/or HBcAb, HBsAb without history of vaccination, human t cell lymphotropic virus 1 (HTLV-1), or hepatitis C virus (HCV)
16. Negative serology for Epstein-Barr virus (EBV) or evidence of acute or chronic infection (IgM ≥ IgG)
17. Lack of updated immunizations per current Centers for Disease Control (CDC) guidelines (including lack of immunization against hepatitis B, pneumococcus and influenza - during season)
18. Presence of panel reactive antibodies > 20%
19. Prostate-specific antigen (PSA) > 4 ng/ml unless malignancy is ruled out
20. Positive tuberculin test (unless proof of adequate treatment for latent tuberculosis can be provided)
21. X-ray evidence of pulmonary infection or other significant pathology
22. Gall stones and/or portal hypertension and/or hemangioma on liver ultrasound
23. Abnormal abdominal or pelvic ultrasound (evidence of masses that are considered suspicious for malignancy or adenopathy)
24. Active peptic ulcer disease
25. Active infections
26. Unstable cardiovascular status (including positive stress echocardiography if age > 35)
27. Untreated or unstable proliferative diabetic retinopathy
28. Previous/concurrent organ transplantation (except for failed islet cell or pancreas transplantation)
29. Malignancy or previous malignancy
30. Any medical condition requiring chronic use of steroids
31. Active alcohol or substance abuse; smoking in the last 6 months.
32. Sexually active females who are not:

    * post-menopausal,
    * surgically sterile, or
    * not using an acceptable method of contraception (oral contraceptives, Norplant, Depo-Provera, and barrier devices with spermicide are acceptable; condoms used alone are not acceptable)
33. Positive pregnancy test or intent for future pregnancy, or male subject's intent to procreate
34. Any condition or any circumstances that make it unsafe to undergo an islet cell transplant
35. Psychogenically unable to comply
36. Failed psychological evaluation
37. Persistent leukopenia (white blood cell count < 3,000/uL on more than 3 occasions)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2005-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, M.D., Principal Investigator — Diabetes Research Institute - University of Miami
Locations (1):
- Diabetes Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Froud T, Baidal DA, Faradji R, Cure P, Mineo D, Selvaggi G, Kenyon NS, Ricordi C, Alejandro R. Islet transplantation with alemtuzumab induction and calcineurin-free maintenance immunosuppression results in improved short- and long-term outcomes. Transplantation. 2008 Dec 27;86(12):1695-701. doi: 10.1097/TP.0b013e31819025e5. PMID 19104407
- [Derived] Tharavanij T, Betancourt A, Messinger S, Cure P, Leitao CB, Baidal DA, Froud T, Ricordi C, Alejandro R. Improved long-term health-related quality of life after islet transplantation. Transplantation. 2008 Nov 15;86(9):1161-7. doi: 10.1097/TP.0b013e31818a7f45. PMID 19005394
- See also: Diabetes Research Institute web site — http://www.diabetesresearch.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Islet Transplantation: Single arm study. Subjects with Type 1 Diabetes, severe hypoglycemia and hypoglycemia unawareness received intrahepatic islet transplantation (1 or 2 infusions) under alemtuzumab induction and rapamycin + MMF maintenance immunosuppression.
Period: Overall Study
Arm/Group | Islet Transplantation
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Glycemic Control by HbA1c and Prevention of Severe Hypoglycemia
Description: Number of subjects at 1 year with HbA1c < 6.5% and absence of severe hypoglycemia
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 3
participants | 3

2. Secondary Outcome: Islet Allograft Function
Description: Number of subjects with basal C-peptide greater than 0.5 ng/ml
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 3
Participants | 3

3. Secondary Outcome: Improvement in Metabolic Control as Evidenced by Hemoglobin A1c < 6.5%
Description: Number of subjects with a hemoglobin A1c < 6.5% at 1year after islet transplantation
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 3
Participants | 3

4. Secondary Outcome: Elimination of Severe Hypoglycemia
Description: The number of subjects with severe hypoglycemia after transplantation
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Restoration of Hypoglycemia Awareness 1 Year After Transplantation
Description: The number of subjects with restoration of hypoglycemia awareness 1 year after islet transplantation
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Islet Transplantation: Islet transplantation alone under alentuzumab (Campath1H) induction.
Arm/Group | Islet Transplantation
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplantation (N=3)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) — lymphopenia secondary to t-cell depletion with alentuzumab (Campath1H)
Hypersensitivity (Immune system disorders) | 1 (1) — chest pain, back pain, abdominal pain with nausea and vomiting after administration of IV iron (Ferrlecit; sodium ferric gluconate) for anemia.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplantation (N=3)
Hair loss (Skin and subcutaneous tissue disorders) | 1 (1)
Displastic Nevus (Skin and subcutaneous tissue disorders) | 1 (1)
Acne/Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Microalbuminuria (Renal and urinary disorders) | 1 (1)
Overt Proteinuria (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Renal and urinary disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (3)
Gallblader polyp (Gastrointestinal disorders) | 1 (1)
Pulpitis (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Right foot injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 (2)
Toe sprain (Musculoskeletal and connective tissue disorders) | 1 (1)
Yeast infection (Reproductive system and breast disorders) | 1 (1)
Uterine fibroids (Reproductive system and breast disorders) | 1 (1)
Hot Flashes (Reproductive system and breast disorders) | 1 (1)
Abnormal Papsmear (Reproductive system and breast disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Tremors (Nervous system disorders) | 1 (1)
Headaches (Nervous system disorders) | 1 (1)
Memory deficit (Nervous system disorders) | 3 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Other (Nervous system disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Edema (Cardiac disorders) | 1 (1)
Thrombophlebitis Right arm (Vascular disorders) | 1 (1)
Capsular opacity (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fatigue (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes